CLINICAL TRIAL: NCT06448104
Title: Effect of Immersive Virtual Reality as a Distraction Tool to Reduce Pain and Discomfort Associated With Dry Needling Application
Brief Title: Virtual Reality in Invasive Techniques in Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3250436
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Pain
Keywords: pain; dry needling; virtual reality
MeSH Terms: conditions — Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry needling and immersive virtual reality (Experimental): Participants assigned to "Dry needling and immersive virtual reality" group will carry out a first session in which the dry needling technique will be performed together with immersive virtual reality and the results will be recorded. Likewise, after two weeks, these participants will repeat the dry needling session (with virtual reality) and evaluation, adding a previous exercise session.
  Interventions: Other: Dry needling and immersive virtual reality
- Standard dry needling (Active Comparator): Participants assigned to "Standard dry needling" group will undergo a first session in which the dry needling technique will be performed and the results will be recorded. After two weeks, these participants will repeat the dry needling and evaluation session, in this case adding a previous exercise session.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling and immersive virtual reality — The study consists of two sessions, separated by a period of two weeks. In the first session, a dry needling procedure based on the Hong technique is performed on the main latent myofascial trigger point of the medial gastrocnemius, vastus medialis quadriceps or biceps femoris muscles.
  The procedure will be carried out simultaneously with the use of immersive virtual reality distraction software, applied through MetaQuest 2 virtual reality glasses. This procedure consists of immersive visualization (video and sound images that represent scenes related to relaxation).
  In the second session, the same procedure will be repeated, with the addition that the participants will perform 3 sets of 10 repetitions (12RM intensity) of the plantar flexion exercises prior to performing the dry needling technique. of ankle, knee extension or knee flexion (depending on the muscle evaluated) with the aim of stimulating the area to be evaluated, simulating post-exercise fatigue.
  Arms: Dry needling and immersive virtual reality
Other: Dry needling — The study consists of two sessions, separated by a period of two weeks. In the first session, a dry needling procedure based on the Hong technique is performed on the main latent myofascial trigger point of the medial gastrocnemius, vastus medialis quadriceps or biceps femoris muscles.
  In the second session, the same procedure will be repeated, with the addition that the participants will perform 3 sets of 10 repetitions (12RM intensity) of the plantar flexion exercises prior to performing the dry needling technique. of ankle, knee extension or knee flexion (depending on the muscle evaluated) with the aim of stimulating the area to be evaluated, simulating post-exercise fatigue.
  Arms: Standard dry needling

SUMMARY:
Dry needling is a common physical therapy technique that uses solid acupuncture needles that are repeatedly inserted and removed into the human body. These techniques, despite their benefits, can cause pain. The objective of this study is to analyze the use of virtual reality as a distractor in invasive techniques in physiotherapy. The hypothesis is that the use of immersive virtual reality, evoking relaxation situations, will reduce the sensation of pain during and/or after the technique. To do this, healthy participants will be recruited and the participants will be divided into two groups (experimental and control). Participants in the experimental group will undergo the dry needling technique on latent myofascial trigger points along with the use of immersive virtual reality. The same technique will be performed on participants in the control group but without the use of virtual reality. Pain during and after puncture and strength after puncture will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one identifiable latent myofascial trigger point in the muscles studied

Exclusion Criteria:

* Suffer any musculoskeletal or neural alteration that could alter the results obtained
* Suffer from belonephobia or extreme and uncontrollable fear of sharp objects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Pain during dry needling | Immediately after technique application in each session (two sessions separated by two weeks)
  Pain perception during dry needling technique measured using a numerical pain rating scale (0-10)

SECONDARY OUTCOMES:
Pain after dry needling | Immediately after technique application; 30 minutes after technique application; 1 hour after technique application; 6 hours after technique application; 24 hours after technique application in each session (two sessions separated by two weeks)
  Pain after dry needling technique measured using a numerical pain rating scale (0-10)
Pain pressure threshold | Before technique; Immediately after technique; 30 minutes after technique; 60 minutes after technique in each session (two sessions separated by two weeks)
  Pain pressure threshold measured using an algometer
Strength | Before technique; Immediately after technique in each session (two sessions separated by two weeks)
  Strength measured using a hand-held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Martín-San Agustín, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy, University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No